CLINICAL TRIAL: NCT05992597
Title: Prospective, Single-arm, Single-center, Phase II Clinical Study of Rituximab, Lenalidomide, Zebutinib Combined Regimen Followed by Sequential Immunochemotherapy in the Treatment of Initially Treated Mantle Cell Lymphoma
Brief Title: ZR2 Sequential Immunochemotherapy for Newly Treated MCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZR2 + RDHAP
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Rituximab, Lenalidomide, Zebutinib ，Mantle Cell Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rituximab, lenalidomide, and zebutinib,RDHAP (Experimental)
  Interventions: Drug: ZR2 RDHAP

INTERVENTIONS:
Drug: ZR2 RDHAP — ZR2:Rituximab 375mg/m2, D1, Lenalidomide 24mg qd D1-14, zebutinib 160mg bid RDHAP:Rituximab 375mg/m2 D0, dexamethasone 40mg D1-4, cytarabine 2g/m2 q12h D2, cisplatin 25mg/m2 D1-3.

SUMMARY:
Patients with newly diagnosed MCL were treated with ZR2 regimen for 3 cycles, followed by 3 cycles of immunochemotherapy, and zebrutinib maintenance therapy for 2 years after the end of induction therapy, in order to improve the remission rate and prognosis of patients with induction therapy.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter, Phase II clinical study evaluating sequential immunochemotherapy followed by rituximab, lenalidomide, and zebutinib combined with or without autologous hematopoietic stem cell transplantation followed by zebutinib maintenance therapy for initial treatment of capsular cell lymphoma. There are three stages: screening, treatment and follow-up. The screening period was 28 days before the first administration. Treatment period: Enrolled subjects first received 3 cycles of rituximab, lenalidomide, zebutinib without chemotherapy (21 days for one cycle), followed by 3 cycles of RDHAP immunochemotherapy (21 days for one cycle); All patients were assessed with interim Positron Emission Tomography (iPET) after 3 cycles of rituximab, lenalidomide, and zebutinib without chemotherapy. All patients will continue to receive 3 cycles Of RDHAP, followed by Treatment End Of Positron Emission Tomography. For patients who have achieved complete metabolic response (CMR) or partial metabolic response (PMR), autologous hematopoietic stem cell transplantation (ASCT) can be performed as consolidation therapy after the researchers evaluate their physical status and their personal wishes. 3 months after ASCT, PET will be reviewed for efficacy evaluation after transplantation. Zebutinib maintenance therapy was started 2 months after transplantation for 2 years. For patients without ASCT, zebutinib maintenance therapy was started directly for 2 years. The follow-up period was entered after the end of maintenance therapy. Efficacy was evaluated using Lugano2014 criteria. Patients with disease progression during non-chemotherapy treatment were directly entered into RDHAP immunochemotherapy, and patients with disease progression during immunochemotherapy were directly removed from the group and entered second-line treatment. Objective effective rate, safety index and survival data of patients were observed during the experiment. Subjects will enter the follow-up period after the study treatment is discontinued or the treatment period has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the clinical study voluntarily: fully understand and be informed of the study and sign the informed consent in person; Willing to follow and be able to complete all test procedures.
* 18~75 years old (inclusive), male and female.
* Histopathologically confirmed mantle cell lymphoma, including positive immunohistochemical CyclinD1 (CyclinD1 or CCND1) and/or chromosomal t (11; 14) (q13; Q32) ectopic.
* No prior anti-tumor therapy, such as chemotherapy, radiotherapy, immunotherapy or biotherapy (tumor vaccine, cytokine, or growth factor controlling cancer).
* there must be at least one evaluable or measurable lesion that meets Lugano2014 criteria (evaluable lesion: PET/CT examination showing increased uptake in lymph nodes or extratodal areas (higher than liver) and PET/CT and/or CT features consistent with lymphoma; Measurable lesions: nodular lesions >15mm in length or extragendal lesions >10mm in length with increased FDG uptake).
* Adequate organ and bone marrow function, no serious hematopoietic dysfunction, abnormal heart, lung, liver, kidney function and immune deficiency (no blood transfusion, granulocytic colony stimulating factor or other relevant medical support within 14 days prior to the use of the study drug) :

A) Blood routine: neutrophil absolute count (ANC) ≥1.5×109/L (1500/mm3), platelet ≥75×109/L, hemoglobin ≥100g/L (if bone marrow is involved, platelet ≥50×109/L, ANC ≥1.0×109/L, hemoglobin ≥80g/L).

B) Liver function: serum bilirubin ≤2.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5 times the upper limit of normal value (AST is allowed if liver is involved, ALT≤5 times the upper limit of normal value).

C) Renal function: creatinine clearance ≥60 mL/min (estimated according to the Cockcroft-Gault formula).

D) Coagulation function: INR≤1.5 times the upper limit of normal value; PT and APTT≤1.5 times the upper limit of normal value.

* Left ventricular ejection fraction (LVEF) ≥ 50% in cardiac function examination.
* Male subjects used effective contraception from signing informed consent until 6 months after the last chemotherapy.
* Life expectancy > 3 months.

Exclusion Criteria:

* The diagnosis was leukemic mantle cell lymphoma.
* Central nervous system involvement secondary to lymphoma.
* history of other active malignant diseases within 2 years prior to study entry, but eligibility for inclusion :(1) adequately treated carcinoma in situ of the cervix; (2) local basal cell carcinoma or squamous cell carcinoma of skin; (3) Pre-existing malignant disease that is under control and has undergone local radical treatment (surgical or other forms).
* People with a known history of Human Immunodeficiency Virus (HIV) infection and/or acquired Immunodeficiency syndrome. Screening stage of hepatitis b surface antigen or hepatitis c virus antibody positive patients, must further by hepatitis b virus DNA (no more than 1000 iu/ml) and HCV RNA detection (shall not exceed the method detection limit), in the activity of the ruled out the need for treatment after hepatitis b or hepatitis c infection, before the experiment. Patients with hepatitis B virus carriers, stabilized hepatitis B after drug treatment and cured hepatitis C can be included.
* Major surgery was performed within 28 days prior to study initiation.
* Any active infections, including but not limited to bacterial, fungal or viral infections, that require systemic antiinfective therapy within 14 days prior to initiation of treatment.
* combined with severe or uncontrolled disease, including but not limited to symptomatic of congestive heart failure, uncontrolled hypertension, unstable angina, active peptic ulcer or A history of severe hemorrhagic diseases, such as hemophilia a., hemophilia B, von willebrand disease or blood transfusion or other medical intervention history of spontaneous bleeding.
* History of stroke or intracranial hemorrhage within 6 months prior to first administration of the study drug.
* A history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months.
* Patients who must take antiplatelet drugs and anticoagulant drugs at the same time due to underlying diseases and have no alternative treatment plan.
* Continuous treatment with strong and moderate CYP3A inhibitors or CYP3A inducers is required. Patients were excluded if they had taken a CYP3A potent or moderate-acting inhibitor or inducer within 7 days prior to the first administration of the study drug (or had taken these drugs for less than 5 half-lives).
* Patients deemed unsuitable for the study by other investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Time Frame: 21days after the end of treatment
  overall response rate

SECONDARY OUTCOMES:
PFS | Time Frame: From date of first day of treatment until the date of first documented progression, assessed up to 24 months
  Progression Free Survival
OS | Time Frame: From date of first day of treatment until the date of first documented date of death from any cause, assessed up to 24 months
  Overall Survival
AE and SAE | Time Frame: From date of first day of treatment until 30 day after last treatment
  Adverse event and serious adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No